CLINICAL TRIAL: NCT03395132
Title: Efficacy and Safety of Fucicort® Lipid Cream Compared to Combination Treatment With Fucidin® Cream Followed by Betamethasone (Lianbang Beisong®) Cream and Fucicort® Lipid Cream Vehicle in Clinically Infected Atopic Dermatitis/Eczema
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to business strategic reasons, LEO Pharma has decided to close down the FCF-38 trial.
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FCF-38
Record Dates: First submitted 2018-01-03; First posted 2018-01-10 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2019-05

CONDITIONS: Infected Atopic Dermatitis/Eczema
MeSH Terms: conditions — Eczema | interventions — Betamethasone

STUDY DESIGN:
Who Masked: Investigator
Masking Description: In order to keep the trial investigator-blind, packaging and labelling of the outer box will be identical for all investigational medicinal products (IMPs). Handling of individual tubes of IMP will therefore be handled by a designated third person. Individual tubes of IMP will be inaccessible for the (sub)investigator and other trial staff involved in evaluation of subjects and conduct of the trial. Subjects will be instructed to only reveal the IMP to the drug dispenser and not to the trial staff.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fucicort® Lipid cream (Experimental): Fucicort® Lipid cream is a combination of the antibiotic fusidic acid (20 mg/g) and the corticosteroid betamethasone (1 mg/g (as 17-valerate)). Twice daily for two weeks.
  Interventions: Drug: Fucicort® Lipid cream
- Fucidin cream +betamethasone cream (Active Comparator): The combination treatment with Fucidin® cream followed by betamethasone (Lianbang Beisong®) cream. Twice daily for two weeks.
  Interventions: Drug: Fucidin® cream; Drug: betamethasone (Lianbang Beisong®) cream
- Vehicle cream (Placebo Comparator): The vehicle cream, also named as Fucicort® Lipid cream vehicle, is the identical cream of Fucicort Lipid cream but without the active ingredient. Twice daily for two weeks.
  Interventions: Drug: Fucicort® Lipid cream vehicle

INTERVENTIONS:
Drug: Fucicort® Lipid cream — The active ingredient of Fucicort® Lipid cream are Fusidic acid and betamethasone. The pack size of Fucicort® Lipid cream is 15g.
  Arms: Fucicort® Lipid cream
Drug: Fucidin® cream — The active ingredient of Fucidin® cream is Fusidic acid. The pack size of Fucidin® cream is 15g.
  Arms: Fucidin cream +betamethasone cream
Drug: Fucicort® Lipid cream vehicle — The active ingredient of Fucicort® Lipid cream vehicle is the identical cream of Fucicort® Lipid cream but without the active ingredient. The pack size of Fucicort® Lipid cream vehicle is 15g.
  Arms: Vehicle cream
Drug: betamethasone (Lianbang Beisong®) cream — The active ingredient of betamethasone (Lianbang Beisong®) cream is Betamethasone hydrate. The pack size of betamethasone (Lianbang Beisong®) cream is 15g.
  Arms: Fucidin cream +betamethasone cream

SUMMARY:
The trial is designed to compare the efficacy and safety of Fucicort® Lipid cream with the combination treatment of Fucidin® cream followed by betamethasone (Lianbang Beisong®) cream, or Fucicort® Lipid cream vehicle, when applied twice daily for two weeks. The trial is designed to demonstrate that treatment with Fucicort® Lipid cream is not inferior to the combination treatment with the mono component drugs, Fucidin® cream followed by betamethasone (Lianbang Beisong®) cream and that treatment with Fucicort® Lipid cream is superior to the treatment with Fucicort® Lipid cream vehicle. This is a 3-arm, parallel group, active- and vehicle-controlled trial comparing the efficacy and safety after 14 days treatment of Fucicort® Lipid cream, to Fucidin® cream followed by betamethasone (Lianbang Beisong®) cream, or Fucicort® Lipid cream vehicle, in subjects with clinically infected AD/eczema.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AD/eczema as defined by Williams's criteria with clinical signs of infected AD/eczema on trunk and/or extremities such as fluid drainage, blistered skin, white or yellow pus, severe itchiness and new burning sensation
* A minimum score of 1 for each of the signs in the m-EASI score in at least one of the pre-defined body areas (trunk and/or extremities)
* Subjects between 2 and 65 years of age

Exclusion Criteria:

* History of concurrent diseases that could interfere with trial assessments or pose a safety concern
* Subjects with other skin lesions, e.g. scarring, tattoos, or hyperpigmentation on the treatment area that could interfere with assessments
* Clinical findings such as severe heart, liver, kidney and lung deficiency, which will be impacted by the trial procedures at the investigator's discretion
* Subjects who have received treatment with any non-marketed drug substance (i.e. an agent which has not yet been made available for clinical use following registration) within the last 4 weeks prior to randomisation at investigator's discretion
* Use of prohibited medication, i.e.

  1. Systemic treatment with immunosuppressive or immunomodulating drugs(including Leigongteng) or corticosteroids within 28 days prior to randomisation
  2. Use of topical or systemic antibiotics and anti-histamines within 14 days prior to randomisation
  3. Phototherapy (e.g. PUVA, UVA or UVB therapy) within 28 days prior to randomisation
  4. Topical treatment with immunomodulators (e.g. pimecrolimus, tacrolimus) within 14 days prior to randomisation
  5. Topical treatment with corticosteroids or any other topical treatment within 7 days prior to randomisation
  6. Use of any non-prescribed systemic or cutaneous medication within 7 days prior to randomisation
  7. The use of analgesics at the discretion of the investigator is allowed before and during the trial

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2019-05-09 (Actual); Study Completion 2019-05-09 (Actual)

PRIMARY OUTCOMES:
The percentage change in modified Eczema Area and Severity Index (m-EASI) on trunk and extremities at Day 15 | from baseline to Day 15
  The percentage change in modified Eczema Area and Severity Index (m-EASI) on trunk and extremities from baseline to Day 15. The m-EASI is a composite score evaluating the severity of 4 clinical signs (erythema, oedema/induration/papulation, excoriation, and lichenification) and the extent of the disease on each of 3 body regions (upper limbs, trunk, and lower limbs) by use of standard scales. The maximum total score is 64.8, with higher values indicating more severe and/or more extensive condition.

SECONDARY OUTCOMES:
Investigator's Global Assessment (IGA) at Day 15 | at Day 15
  The IGA of disease severity on the body (trunk and extremities, excluding the hands, head, and neck) will be assessed based on a visual evaluation by use of definitions of severity ranging from 0 (clear) to 5 (very severe).
Controlled disease according to IGA | at Day 15
  Controlled disease according to IGA at Day 15, defined as subjects having at least 'moderate' disease at baseline achieving 'clear' or 'almost clear' disease severity or subjects having 'mild' disease at baseline achieving 'clear' according to IGA.
Proportion of patients with successful bacteriological response | at Day 15
  Proportion of patients with successful bacteriological response, defined as pathogens present on target lesion at baseline and either: a) no pathogen present on target lesion at Day 15 ('confirmed eradication') or b) no swab taken at Day 15 as no lesion was evident ('presumptive eradication').
Adverse event (AE)/serious adverse event (SAE) frequency | baseline to Day 15 and 14±2 days follow up or until the final outcome is determined
  Adverse event (AE)/serious adverse event (SAE) frequency by preferred term. Ongoing (serious or non-serious) AE with a possible, probable, or non-assessable relationship to the IMP at the last visit in the treatment phase. The investigator should follow up on the outcome for 14±2 days or until the final outcome is determined. This follow-up visit can be made either as a phone call or as a regular visit according to the investigator's discretion.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — LEO Pharma
Locations (15):
- China (15):
  - Beijing Children's Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Guangdong General Hospital, Guangzhou, Guangzhou
  - Tongji Hospital of Tongji Medical College of Huazhong Univ. of Science & Technology, Wuhan, Hubei
  - Dermatology Hospital, China Academy of Medicine and Science, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Hospital of Dalian Medical University, Dalian, Liaoning
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - The Chinese People's Liberation Army General Hospital Of Northern Theater, Shenyang, Liaoning
  - The People's Hospital of Liaoning Province, Shenyang, Liaoning
  - Tangdu Hospital, Xi'an, Shan'xi
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Shanghai Huashan Hospital, Shanghai, Shanghai Municipality
  - Children's Hospital of Shanghai, Shanghai, Shanghai Municipality
  - Children's Hospital, Capital Institute of Pediatrics, Beijing

IPD SHARING:
Plan to Share IPD: No